CLINICAL TRIAL: NCT06863805
Title: Evaluation of the Clinical Utility of Circulating Biomarkers in Advanced Thyroid Carcinomas
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: BIOTYR; RC-2022-2773340 (Other Grant/Funding Number: IRCCS Azienda Ospedaliero universitaria Bologna)
Record Dates: First submitted 2025-01-10; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-11

CONDITIONS: Thyroid Carcinoma
Keywords: carcinomas of thyroid; molecular markers; liquid biopsy
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with advanced thyroid carcinomas: Adults patients with advanced thyroid carcinomas will be enrolled.
  Interventions: Diagnostic Test: 4 EDTA tubes of peripheral blood for Multigene analysis on ccf-DNA and ccf-RNA

INTERVENTIONS:
Diagnostic Test: 4 EDTA tubes of peripheral blood for Multigene analysis on ccf-DNA and ccf-RNA — For each patient enrolled in the present study, 4 EDTA tubes of peripheral blood will be collected to be used to obtain molecular profiling during scheduled laboratory controls as per normal clinical practice according to the following time schedule:
  * T0 = basal collection before initiation of systemic treatment;
  * T1 = sampling at 1 month after the start of systemic treatment;
  * T2 = sampling at 3 months (+/- 1 month) after the start of systemic treatment at the first instrumental re-evaluation of disease;
  * T3 = sampling at 6 months (+/- 1 month) from the start of systemic treatment at the time of instrumental disease reassessment;
  * T4 = sampling at the time of evidence of instrumental disease progression within 24 months of treatment initiation.
  The following analyses will be conducted on the samples thus collected:
  * multigenic analysis on ccf-DNA and ccf-RNA at baseline, i.e., before the initiation of systemic treatment;
  * isolation, counting and analysis of CTCs at baseline vi

SUMMARY:
The study is aimed at all adult patients diagnosed with advanced thyroid carcinomas and well-differentiated thyroid carcinomas (DTC) iodine-refractory, well-differentiated iodine-refractory thyroid (RAI-R DTC) metastatic carcinomas that are candidates for systemic therapy. By simple blood sampling and analysis on peripheral blood of circulating DNA (ccf-DNA), circulating RNA (ccf-RNA), and counting and analysis of circulating tumor cells through the use of liquid biopsy, molecular profiling corresponding to those obtained by genomic sequencing on tumor tissue can be arrived at, depending on optimal therapeutic choices

DETAILED DESCRIPTION:
In recent years, research has focused on the so-called "liquid biopsy," understood as a noninvasive procedure capable of performing analysis on tumor-derived material contained in blood such as circulating free DNA (ccf-DNA), circulating free RNA (ccf-RNA), and circulating tumor cells (CTCs), capable of providing a dynamic snapshot of the molecular structure of the oncological pathology throughout its course.

In thyroid cancers, liquid biopsy methods have also proven feasible with potential clinical applications, both in the prognostic field, in the identification and monitoring of minimal residual disease, and in therapeutics. 28 The identification, in fact, of circulating biomarkers predictive of response or resistance to drugs in use to date first and foremost would allow in clinical practice a more accurate selection of patients at the time of initiation of systemic treatment, especially where tumor tissue is not available or adequate for molecular profiling. In addition, the identification of new molecular events, even secondary ones, during treatment would offer the possibility of developing alternative therapeutic strategies aimed at overcoming resistance.

The primary objective of the present study is to verify the match between molecular profiling obtained by liquid biopsy versus that obtained by genomic sequencing on tumor tissue (gold standard) in patients with advanced thyroid carcinoma who are candidates for systemic therapy.

The secondary objectives of this study are as follows:

* identification of circulating biomarkers predictive of response to cancer treatment useful for selecting patients with iodine-resistant metastatic disease for initiation of systemic therapy by profiling on peripheral blood;
* identification of additional molecular events, expression of polyclonal disease evolution, that may represent new therapeutic targets.

The study is interventional low-risk, tissue-based, prospective, single-center study.

For each patient enrolled in the present study, 4 EDTA tubes of peripheral blood will be collected to be used to obtain molecular profiling during scheduled laboratory controls as per normal clinical practice according to the following time schedule:

* T0 = basal collection before initiation of systemic treatment;
* T1 = sampling at 1 month after the start of systemic treatment;
* T2 = sampling at 3 months (+/- 1 month) after the start of systemic treatment at the first instrumental re-evaluation of disease;
* T3 = sampling at 6 months (+/- 1 month) from the start of systemic treatment at the time of instrumental disease reassessment;
* T4 = sampling at the time of evidence of instrumental disease progression within 24 months of treatment initiation.

The following analyses will be conducted on the samples thus collected:

* multigenic analysis on ccf-DNA and ccf-RNA at baseline, i.e., before the initiation of systemic treatment;
* isolation, counting and analysis of CTCs at baseline visit
* multigenic analysis on ccf-DNA and ccf-RNA and isolation, counting and analysis of CTCs during treatment (at + 1 month, + 3 months, + 6 months and at progression)
* Outcome of the primary study objective: presence of gene alterations (BRAF mutations, RAS mutations, RET mutations, rearrangements of NTRK, RET, ALK, etc.) found in the two molecular profiling methods, performed on peripheral blood and tumor tissue.
* Outcome of the study secondary objectives: early metabolic response rate assessed by fluorodeoxyglucose (FDG) CT-PET at one month of treatment; overall response rate (ORR); progression-free survival (PFS); tumor burden assessed by sum of diameters (SOD) of measurable disease according to RECIST v.1.1 criteria; isolation, count (CTC/ml) and phenotype assessment of CTCs.

The results obtained will be compared with those obtained from biomolecular profiling of disease on tumor tissue that is already available as per clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent,
* Adult (≥18 years) male or female patients
* Histologic diagnosis of advanced thyroid carcinoma confirmed at centralized review,
* well-differentiated thyroid carcinomas, medullary thyroid carcinomas, anaplastic thyroid carcinomas, advanced, candidates for initiation of systemic medical therapy,
* Availability of biomolecular profiling performed by multigenic NGS panel on tumor tissue,
* Measurable disease by conventional imaging adopted in clinical practice (total body CT with mdc, CT-PET with FDG or F-DOPA).

Exclusion Criteria:

* Patients already receiving previous lines of systemic therapy,
* Patients not eligible for systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients (≥ 18 years) with metastatic RAI-R DTC who are candidates for systemic therapy, as per clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Genomic alterations | Before the start of pharmacologic treatment and after 30 days and 3, 6 and 24 months after the start of treatment
  Presence of BRAF mutations, RAS mutations, RET mutations, rearrangements of NTRK, RET, ALK, etc. in ccf-DNA, ccf-RNA and Circulating Tumour Cells (CTCs)

SECONDARY OUTCOMES:
Early metabolic response rate | 30 days from the start of pharmacologic treatment
  Early metabolic response rate evaluated by FDG-PET
Overall response rate (ORR) | Throughout the study duration, an average of 24 months
  Rate of clinical response
Progression-free survival (PFS) | Throughout the study duration, an average of 24 months
  Progression-free survival (PFS) assessed throughout the study
Tumour load | Throughout the study duration, an average of 24 months
  Calculated as sum of diameters (SOD) of measurable disease according to RECIST v.1.1 criteria
Number of Circulatin Tumour cells (CTC) (CTC/ml) | Before the start of pharmacologic treatment and after 30 days and 3, 6 and 24 months after the start of treatment
  CTC number expressed as CTC/ml
Circulatin Tumour Cells phenotype | Before the start of pharmacologic treatment and after 30 days and 3, 6 and 24 months after the start of treatment
  Description of the CTC phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Ianni, Study Chair — Ospedale S. Orsola-Malpighi
Locations (1):
- IRCCS Azienda Ospedaliero universitaria Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No